CLINICAL TRIAL: NCT03461822
Title: Study of Effectiveness of Stereotactic Body RadioTherapy and Stereotactic RadioSurgery in Solid Primary Inoperable and Oligometastatic Cancer
Brief Title: Effectiveness of Stereotactic RadioTherapy in Solid Primary Inoperable and Oligometastatic Cancer
Acronym: ESRTSPIOC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The National Center of Oncology, Azerbaijan (Other Government)
Responsible Party: Principal Investigator, Azer Aliyev, Radiation Oncologist, PhD, The National Center of Oncology, Azerbaijan
Other Study IDs: MOM-0005
Record Dates: First submitted 2018-02-20; First posted 2018-03-12 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Radiotherapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- SRT in primary-inoperable solid tumors: stereotactic radiotherapy in hypofractionated regimes in 1-5 fractions in primary-inoperable solid tumors
- Classic radiotherapy in primary-inoperable solid tumors: Classic radiotherapy in 1.8-2.0 Gy per fraction in primary-inoperable solid tumors
- SRT in oligometastatic cancer: stereotactic radiotherapy in hypofractionated regimes in 1-5 fractions in oligometastatic cancer
- Classic radiotherapy in oligometastatic cancer: Classic radiotherapy in 1.8-2.0 Gy per fraction in oligometastatic cancer

SUMMARY:
The purpose of this study is to development of more effective treatment tactics of the stereotactic radiotherapy and radiosurgery alone and together with classic radiation therapy in primary inoperabel solid tumors and oligometastastatic cancer.

DETAILED DESCRIPTION:
Despite the fact that of many investigations in the world clinical researches, the SRT of primary-inoperabel and metastatic solid tumors combined with conventional and conformal radiation therapy methods the possibility of the sequences, the optimal fractions of the regimes and doses which determines normal tissues toxic manifestations, implementation of prevention, have not been solved yet.

The conducted research works to study quality of life for improving the social status of patients with primary-inoperable and metastatic solid tumors, is not fully resolved.

Thus, preparing of highly effective treatment tactics in primary-inoperable and metastatic solid tumors, is one of the most important problems of modern clinical oncology and this fact gives grounds to carry out the planned research work.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary-inoperable solid tumors or oligometastatic cancer.
* Acceptance of patient by surgeon as non-operabel or refusing of surgery.
* No more than 4 metastatic foci in irradiated organ.
* Karnofsky scale more than 60.
* Age ≥18 years.
* Estimated duration of life >3 months.
* Hemoglobin ≥ 8 g/dl.
* Absolute neutrophil count at least 1,500/mm^3.
* Platelet count at least 70,000/mm^3.
* Bilirubin no greater than 1.5 times normal.
* SGOT and SGPT no greater than 3 times normal.
* Creatinine less than 1.5 mg/dL. PT-INR/APTT less than 1.5.
* Last patients data no older than 1 month.
* No prior radiotherapy of same location.
* Prior chemottherapy more than 2 weeks ago.

Exclusion Criteria:

* Progression of primary site of metastatic cancer.
* Pregnancy or Breast-Feeding.
* Decompensated concomitant diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The groups will be selected from patients which referred to National Center of Oncology and matching for conducting radiotherapy and Eligibility Criteria.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2013-03; Primary Completion 2019-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Relapse Rate (local and/or distant) | 5 years
  clinical-instrumental or laboratory signs of local and/or distant recurrences of previously diagnosed oncological diaseases
Number of Deaths Due to Any Cause | 5 years
  Deaths due to any complications or progression of previously diagnosed oncological diaseases

SECONDARY OUTCOMES:
Incidence of acute toxicity | Up to 90 days after completion of radiation therapy
  Number of adverse effects of irradiation observed in the patients within 3 months from the begginning of the treatment, measured by CTCAE 4.03 and/or EORTC/RTOG scales.
Incidence of late toxicity | Up to 2 years after completion of radiation therapy
  Number of adverse effects of irradiation observed in the patients after 3 months from the begginning of the treatment, measured by LENT SOMA scale.

CONTACTS AND LOCATIONS:
Locations (1):
- National Center of Oncology, Baku, Azerbaijan

IPD SHARING:
Plan to Share IPD: No